CLINICAL TRIAL: NCT05547646
Title: The Prevalence of Healthcare-associated Infection in Medical Intensive Care Units in Tunisia: NOSOREA2 Study
Brief Title: The Prevalence of Healthcare-associated Infection in Medical Intensive Care Units in Tunisia
Acronym: NOSOREA2
Status: Completed | Type: Observational
Sponsor: Abderrahmane Mami Hospital (Other)
Responsible Party: Principal Investigator, Amira JAMOUSSI, Dr Associate Professor, Abderrahmane Mami Hospital
Other Study IDs: 1
Record Dates: First submitted 2022-09-01; First posted 2022-09-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Cross Infection; Prevalence; Epidemiology; Critical Care
Keywords: Iatrogenic Disease; Cross Infection; Intensive Care Units; Prevalence; Risk Factors; Critical Care
MeSH Terms: conditions — Cross Infection; Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aimed to determine the prevalence of HAI in medical Tunisian ICUs. Secondary endpoints were to identify the predominant infecting microorganisms and evaluate independent risk factors of HAIs.

DETAILED DESCRIPTION:
In Tunisia, there is no national or regional monitoring system of HAI. It is worth noting that HCAIs in intensive care unit (ICU) are more common and life threatening than in general ward because of the frequent use of invasive procedures and multiple therapies.

Controlling this fatal scourge should begin with greater awareness of HAI frequency and ICU ecology. That is why conducting multi-center Tunisian studies is necessary to guide control measurements against HAI and to improve surveillance and infection-control practices. NOSOREA1 study (Tunis Med. 2018 Oct-Nov;96(10-11):731-736) was conducted in 2017 and showed that HAI prevalence within Tunisian ICUs was 25.2% CI 95% [15-35]. Five years later, it is high time to update our finding.

ELIGIBILITY:
Inclusion Criteria:

* All patients occupying an ICU bed over a 48-hour period
* Age >=18 years

Exclusion Criteria:

* no criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One-day point-prevalence study (September 27th, 2022) All medical ICUs across Tunisia are invited to participate, excluding cardiologic and paediatric care units.
  All patients occupying an ICU bed over a 48-hour period are eligible.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Determine the prevalence of healthcare-associated infection in medical Tunisian ICUs | September 27th, 2022
  The number of infected patients divided by the total number of patients at the day of the study

SECONDARY OUTCOMES:
Identify independent risk factors of HAIs. | September 27th, 2022
  Multivariate logistic regression model

CONTACTS AND LOCATIONS:
Overall Officials: Amira JAMOUSSI, pROFESSOR, Principal Investigator — Ministery of Health
Locations (1):
- Medical ICU, Tunis, Ariana Governorate, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided